CLINICAL TRIAL: NCT01237145
Title: Study to Determine the Immune Response From Broncho-alveolar Cells Against Pigeon Specific Antigens
Brief Title: Bronchoalveolar Immune Response Determination
Acronym: BIRD
Status: Completed | Type: Observational
Sponsor: Bossink, A.W.J. (Individual)
Responsible Party: Principal Investigator, A.W.J.Bossink, Dr, Bossink, A.W.J.
Other Study IDs: BIRD01
Record Dates: First submitted 2010-11-07; First posted 2010-11-09 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Extrinsic Allergic Alveolitis
Keywords: pigeon; bird fancier; extrinsic allergic alveolitis; BAL; broncho-alveolar lavage; elispot; antigen
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cells obtained from Broncho alveolar lavage and blood collection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- non-EAA, pigeon: subject with BAL because of diseases not suspected to be EAA
- EAA, pigeon: Bird fanciers with a typical clinical presentation suspected for pigeon induced EAA

SUMMARY:
The purpose of this study is to establish if cells present in lung tissue during extrinsic allergic alveolitis (EAA) are able to elicit an immune response against specific antigens. The hypothesis is: cells in BAL lavage fluid from patients with EAA will be responsive to specific antigens and this response can be measured using ELISPOT.

DETAILED DESCRIPTION:
Subjects suffering from extrinsic allergic alveolitis caused by pigeons will undergo a broncho alveolar lavage. Cells obtained from this BAL will be used for ELISPOT technique with pigeon specific antigens

ELIGIBILITY:
Inclusion Criteria:

* suspicion of pigeon induced extrinsic alveolitis

Exclusion Criteria:

* use of oral steroids
* unable to give informed consent
* age below 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected to have pigeon induced extrinsic allergic alveolitis will be recruited by advertisment in bird fanciers journals. Controls will be patients at the department of pulmonology and tuberculosis needing examination for other reasons
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
ELISPOT response in cells obtained from broncho-alveolar lavage | 2 days
  All elispots will be performed the same day, the end point will be available the next day

SECONDARY OUTCOMES:
Elispot response in cells from blood | 2 days
  ELispots will be performed the same day as blood collection, results will be available the next day

CONTACTS AND LOCATIONS:
Overall Officials: Aik Bossink, MD PhD, Principal Investigator — Diakonessenhuis, Utrecht
Locations (1):
- Diakonessenhuis Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Jafari C, Thijsen S, Sotgiu G, Goletti D, Dominguez Benitez JA, Losi M, Eberhardt R, Kirsten D, Kalsdorf B, Bossink A, Latorre I, Migliori GB, Strassburg A, Winteroll S, Greinert U, Richeldi L, Ernst M, Lange C; Tuberculosis Network European Trialsgroup. Bronchoalveolar lavage enzyme-linked immunospot for a rapid diagnosis of tuberculosis: a Tuberculosis Network European Trialsgroup study. Am J Respir Crit Care Med. 2009 Oct 1;180(7):666-73. doi: 10.1164/rccm.200904-0557OC. Epub 2009 Jul 9. PMID 19590020
- [Background] Losi M, Bossink A, Codecasa L, Jafari C, Ernst M, Thijsen S, Cirillo D, Ferrarese M, Greinert U, Fabbri LM, Richeldi L, Lange C; European Tuberculosis Network TBNET. Use of a T-cell interferon-gamma release assay for the diagnosis of tuberculous pleurisy. Eur Respir J. 2007 Dec;30(6):1173-9. doi: 10.1183/09031936.00067307. Epub 2007 Aug 22. PMID 17715165
- [Background] Kosters K, Nau R, Bossink A, Greiffendorf I, Jentsch M, Ernst M, Thijsen S, Hinks T, Lalvani A, Lange C. Rapid diagnosis of CNS tuberculosis by a T-cell interferon-gamma release assay on cerebrospinal fluid mononuclear cells. Infection. 2008 Dec;36(6):597-600. doi: 10.1007/s15010-007-7316-0. Epub 2008 Jan 12. PMID 18193383